CLINICAL TRIAL: NCT04714515
Title: Using Montelukast to Treat the Patients Infected With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Brief Title: Montelukast - a Treatment Choice for COVID-19
Status: Completed | Type: Observational
Sponsor: University of Sargodha (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other); Shanghai Jiao Tong University School of Medicine (Other); Teesside University (Other)
Responsible Party: Principal Investigator, Muhammad Fayyaz ur Rehman, Principal Investigator, University of Sargodha
Other Study IDs: 01032020-7
Record Dates: First submitted 2020-09-19; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: COVID-19; Montelukast
MeSH Terms: conditions — COVID-19 | interventions — montelukast; Hydroxychloroquine; Ivermectin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Nasal Swab samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (4):
- Hydroxychloroquine and Montelukast: Group 1 was given Standard of care (SOC) + HCQ + Montelukast
  Interventions: Drug: Montelukast; Drug: Hydroxychloroquine
- Montelukast: Group 2 was given Standard of care (SOC) + Montelukast
  Interventions: Drug: Montelukast
- Hydroxychloroquine: Group 3 was given Standard of care (SOC) + HCQ
  Interventions: Drug: Hydroxychloroquine
- Hydroxychloroquine, Montelukast and Invermectin: Group 4 was given Standard of care (SOC) + Montelukast + HCQ and Ivermectin
  Interventions: Drug: Montelukast; Drug: Hydroxychloroquine; Drug: Ivermectin

INTERVENTIONS:
Drug: Montelukast — An FDA approved medicine to treat asthmatic patients
  Groups: Hydroxychloroquine and Montelukast; Hydroxychloroquine, Montelukast and Invermectin; Montelukast
Drug: Hydroxychloroquine — An FDA approved antiarthritis drug
  Groups: Hydroxychloroquine; Hydroxychloroquine and Montelukast; Hydroxychloroquine, Montelukast and Invermectin
Drug: Ivermectin — An FDA approved anti-parasitic medicine
  Groups: Hydroxychloroquine, Montelukast and Invermectin

SUMMARY:
The current study aimed to make a therapeutic comparison and effectiveness of Hydroxychloroquine (HCQ) and Montelukast (ML) in COVID-19 patients in addition to the standard of care. The safety and efficacy of HCQ and ML will be assessed as individual therapy and in combination with each other and with the standard of care. Cytokine storm (Interleukin levels) also will be monitored throughout the study to assess treatment progression.

DETAILED DESCRIPTION:
To date, no specific medication is available for COVID-19. Many FDA-approved drugs, including antivirals, antibacterials, and anti-inflammatory compositions are being tested with the intention of repurposing against COVID-19. In this study, investigators have evaluated the effectiveness of Hydroxychloroquine (HCQ) and Montelukast (ML) in an individual and combination therapy.

Investigators have performed an observational study of 100 hospitalized COVID-19 patients while assessing the safety and efficacy of HCQ, ML, and IV as individual therapy and in combination with each other. ECG, interleukin levels, LFTs, blood profiles were continuously monitored throughout the study.

The aim was to observe participants treated with ML and monitor the inflammatory markers to see whether they increase or decrease and whether an increase in survival rate is observed. The findings have shown that combinational therapy of ML with continuous observation of liver/kidney profiles and QTc prolongation can provide robust recovery with suppression of cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed COVID-19
* Patients who are not directly admitted to ICU

Exclusion Criteria:

* Patients, who were already on immunosuppressants
* Patients with age > 80
* Patient with any known allergies to montelukast

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who were admitted to the hospitals with SARS-CoV-2 contacts (environmental exposure or close contact) or obvious COVID-19 symptoms and were diagnosed with COVID-19 using the PCR tests. Consent was obtained from all patients with a detailed history of any known co-morbidities.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Patients admittance to ICU | 2 Week
  Changes in the number of ICU visits of COVID-19 patients
Length of total stay at the hospital | 2 weeks
  Changes in the length of total stay of patients at the hospital
Alleviating the symptoms of COVID-19 | 2 weeks
  Monitoring the changes in disease severity with alleviation of the symptoms

SECONDARY OUTCOMES:
Interleukin levels | 1 Week
  Monitoring the Interleukin levels with the progression of treatments

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, MD, Principal Investigator — Department of Critical Care Medicine, Shanghai General Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China; Muhammad Rehman Akram, MBBS, Principal Investigator — Shaukat Khanum Memorial Cancer Hospital & Research Centre, Johar Town, Lahore, Pakistan
Locations (2):
- Department of Critical Care Medicine, Shanghai General Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China, Shanghai, China
- Shaukat Khanum Memorial Cancer Hospital & Research Centre, Johar Town, Lahore, Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided